CLINICAL TRIAL: NCT00501982
Title: An International, Open, Randomized, Controlled Study to Evaluate the Efficacy of Combining Prophylactic Curosurf® With Early Nasal CPAP Versus Early Nasal CPAP Alone in Very Preterm Infants at Risk of Respiratory Distress Syndrome
Brief Title: Efficacy of Combining Prophylactic Curosurf With Early Nasal CPAP in Delivery Room: the Curpap Study
Acronym: Curpap
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: DM/PR/5000/002/04
Record Dates: First submitted 2007-07-16; First posted 2007-07-17 (Estimated); Last update posted 2020-08-03 (Actual); Status verified 2020-07

CONDITIONS: Respiratory Distress Syndrome, Newborn
Keywords: surfactant; RDS; nCPAP; Mechanical Ventilation; Premature Infants; Neonatal Respiratory Distress Syndrome (nRDS)
MeSH Terms: conditions — Respiratory Distress Syndrome, Newborn; Premature Birth | interventions — poractant alfa

ARMS (2):
- 1 (No Intervention): N Cpap in delivery room and than rescue curosurf in case of need
- 2 (Experimental): Poractant alfa (Curosurf) + N Cpap in delivery room
  Interventions: Drug: Poractant alfa (Curosurf®)

INTERVENTIONS:
Drug: Poractant alfa (Curosurf®)
  Arms: 2

SUMMARY:
The primary objective of this study is to compare two methods of post-delivery stabilization and subsequent early respiratory care for reducing the need for MV and related secondary complications, such as BPD, in premature babies at high risk of RDS:

1. Early stabilization on nCPAP
2. Intubation, prophylactic surfactant (Curosurf®) administration shortly after delivery, and rapid extubation to nCPAP.

The data obtained from this comparison will be applied to test the hypothesis that preterm neonates at risk of RDS who are treated with prophylactic surfactant + nCPAP show less need for MV when compared to infants who receive nCPAP alone.

ELIGIBILITY:
Inclusion Criteria:

* Preterm neonates with a gestational age (GA) of 25+0 - 28+6 completed weeks.
* Inborn neonates.
* In case of twins, both neonates will be included in the same treatment arm.
* Parental written informed consent for participation in the study obtained on admission into the hospital or prior to delivery.

Exclusion Criteria:

* Evidence of severe birth asphyxia, that is an APGAR score below 3 at 5 minutes of age.
* Need for endotracheal intubation for cardiopulmonary resuscitation or insufficient respiratory drive.
* Known genetic or chromosomal disorders.
* Delivered to mothers with ruptured membranes of more than 3 weeks duration.
* Potentially life-threatening conditions unrelated to immaturity.
* Participation in another clinical trial of any placebo, drug, biological, or device conducted under the provisions of a protocol.

Ages: 25 Weeks to 28 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 208 (Actual)
Dates: Start 2007-03; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Need for MV | Within the first 5 days of life

SECONDARY OUTCOMES:
Incidence of BPD and other complications of prematurity. Lenght of hospitalization. Clinical status until discharge home | entire study

CONTACTS AND LOCATIONS:
Overall Officials: Laura Fabbri, Study Director — Medical Department; Chiesi Farmaceutici S.p.A (Italy)
Locations (5):
- General Faculty Hospital, Prague, Czechia
- Hopital De La Conception, Marseille, France
- Ospedale Maggiore, Bologna, Italy
- Maternidade Alfredo da Costa, Lisbon, Portugal
- Hospital De Cruces, Bilbao, Spain

REFERENCES:
- [Result] Sandri F, Plavka R, Ancora G, Simeoni U, Stranak Z, Martinelli S, Mosca F, Nona J, Thomson M, Verder H, Fabbri L, Halliday H; CURPAP Study Group. Prophylactic or early selective surfactant combined with nCPAP in very preterm infants. Pediatrics. 2010 Jun;125(6):e1402-9. doi: 10.1542/peds.2009-2131. Epub 2010 May 3. PMID 20439601
- See also: Study Record on EU Clinical Trials Register including results — https://www.clinicaltrialsregister.eu/ctr-search/search?query=2006-004105-25